CLINICAL TRIAL: NCT02230202
Title: Endothelial Microparticles: A Novel Marker of Vascular Dysfunction
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1209; UL1TR001082 (NIH)
Record Dates: First submitted 2014-08-25; First posted 2014-09-03 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — plasma and urine biospecimens to be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy control: Healthy control that meets inclusion/exclusion criteria. Single blood draw and flow-mediated dilation (FMD).
  Interventions: Other: Flow-mediated dilation; Other: single blood draw
- Stage III or IV CKD patients: Stage III or IV CKD patients that meets inclusion/exclusion criteria. Single blood draw and flow-mediated dilation (FMD).
  Interventions: Other: Flow-mediated dilation; Other: single blood draw
- Post-transplant patients: Stage III or IV CKD Post-transplant patients that meets inclusion/exclusion criteria. Single blood draw and flow-mediated dilation (FMD).
  Interventions: Other: Flow-mediated dilation; Other: single blood draw

INTERVENTIONS:
Other: Flow-mediated dilation — Flow-mediated dilation used to measure vascular function. The test is minimally invasive, with only a slight discomfort due to the inflation of the arm cuff.
Other: single blood draw — single blood draw of approximately 45 mL.

SUMMARY:
The primary hypothesis of this proposal is that chronic kidney disease (CKD) and treatment with calcineurin inhibitors (CNIs) are each associated with the release of endothelial microparticles into the plasma.

DETAILED DESCRIPTION:
The primary hypothesis of this proposal is that chronic kidney disease (CKD) and treatment with calcineurin inhibitors (CNIs) are each associated with the release of endothelial microparticles into the plasma. These injury-associated microparticles have a different molecular/protein composition than those released from endothelial cells in healthy patients, and their abundance correlates with vascular injury. To test this hypothesis the investigators propose a 3 arm case-controlled study including normal controls, individuals with stage III and IV CKD not receiving CNI therapy, and individuals with stage III and IV CKD post kidney transplantation receiving a CNI. The goal of this study is to measure the amount of microparticles in patients with kidney disease who have had a kidney transplant. Another goal of this study is to see if the measurements of microparticles are related to poor function of the vessels (endothelial dysfunction).

ELIGIBILITY:
Inclusion Criteria:

For Healthy controls:

* BMI less than 40 kg/m^2
* Able to give informed consent

For Stage III or IV CKD patients:

* BMI less than 40 kg/m^2
* Able to give informed consent
* An estimated Glomerular-Filtration Rate (GFR) of 20-60 mL/min/1.73m^2

For Post-kidney transplant and stage III or IV CKD patients:

* BMI less than 40 kg/m^2
* Able to give informed consent
* An estimated Glomerular-Filtration Rate (GFR) of 20-60 mL/min/1.73m^2

Exclusion Criteria:

For Healthy controls:

-Women pregnant or breastfeeding

For Stage III or IV CKD patients:

* Women pregnant or breastfeeding
* Adults with a life expectancy of less than one year
* A history of significant liver disease or congestive heart failure
* Hospitalization within the last three months
* Active infection on antibiotic therapy
* Uncontrolled hypertension (>140/90)
* Immunosuppressive therapy within the last year

For Post-transplant stage III or IV CKD patients:

* Women pregnant or breastfeeding
* Adults with a life expectancy of less than one year
* A history of significant liver disease or congestive heart failure
* Hospitalization within the last three months
* Active infection on antibiotic therapy
* Uncontrolled hypertension (>140/90)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90 volunteers from the Anschutz Medical Campus
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Vascular Function | percent change from baseline over 2 minutes
  This will be measured with flow-mediated dilation and evaluate percent change from baseline over minutes.

SECONDARY OUTCOMES:
Characterization of Microparticle source from blood analysis | Single time point
  A single blood draw to distinguish micro particle source characterization based upon protein, lipid and cholesterol composition.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Thurman, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus; CTRC, Aurora, Colorado
  - University of Colorado School of Medicine, Aurora, Colorado

REFERENCES:
- [Derived] Jalal D, Renner B, Laskowski J, Stites E, Cooper J, Valente K, You Z, Perrenoud L, Le Quintrec M, Muhamed I, Christians U, Klawitter J, Lindorfer MA, Taylor RP, Holers VM, Thurman JM. Endothelial Microparticles and Systemic Complement Activation in Patients With Chronic Kidney Disease. J Am Heart Assoc. 2018 Jul 13;7(14):e007818. doi: 10.1161/JAHA.117.007818. PMID 30006493